CLINICAL TRIAL: NCT04574466
Title: Scaling-up Psychological Interventions With Syrian Refugees in Switzerland: RCT
Brief Title: Scaling-up Psychological Interventions With Syrian Refugees in Switzerland (STRENGTHS_CH): RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BASEC-2017-01175-rct
Record Dates: First submitted 2020-09-16; First posted 2020-10-05 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Distress; PTSD; Anxiety; Depression; Trauma; Functional Disabilities; Common Mental Health Problems
Keywords: Problem Management Plus; Distress; Mental Health Care; Low-intensity; Refugees
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The definitive RCT will inform us about the effectiveness and implementation of the intervention.
  After the baseline assessment, three hundred eighty participants (N = 380) will be involved in the exploratory RCT (assigned to either the PM+ intervention (n=190) or the ETAU control condition (n=190)).
Who Masked: Outcomes Assessor
Masking Description: All instruments and questions will be administered using tablets by trained research staff blind to the allocation status of the participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Treatment As Usual (ETAU) (No Intervention): The control group will receive enhanced treatment as usual (ETAU). ETAU means that the research team will advise the participants to contact their doctor in case of physical or mental health problems. Moreover, the research team will hand over written information (official booklet) about the operating of the Swiss health care system. Adequate treatment will be provided by a physician, usually, a general practitioner who acts as a gate-keeper (an asylum seeker or refugee has to go first to his/her assigned GP in order to get access to the health care system).
- Problem Management Plus (Experimental): The participants who are assigned to the intervention group will receive five sessions of PM+, a psychological intervention which has been developed by the WHO. PM+ is a new short, transdiagnostic (i.e., not specifically aimed at treating a certain mental disorder) program aiming to reduce common mental health symptoms and improve psychosocial functioning.
  PM+ is a new, brief, psychological intervention program based on Cognitive Behaviour Therapy (CBT) techniques that are empirically supported and formally recommended by the WHO. The full protocol was developed by the WHO and the University of New South Wales, Australia. The manual involves the following empirically supported elements: problem solving plus stress management, behavioural activation, and accessing social support. These elements have been recommended in recent WHO guidelines. PM+ has proven to be effective by two randomized controlled trials (RCTs) in Kenya and Pakistan.
  Interventions: Behavioral: Problem Management Plus

INTERVENTIONS:
Behavioral: Problem Management Plus — Problem Management Plus (PM+) is a new, brief, psychological intervention program based on CBT techniques that are empirically supported and formally recommended by the WHO. The full protocol was developed by the WHO and the University of New South Wales, Australia. The manual involves the following empirically supported elements: problem solving plus stress management, behavioural activation, facing fears, and accessing social support. These elements have been recommended in recent WHO guidelines.
  Arms: Problem Management Plus

SUMMARY:
The current refugee crisis across the Middle East and Europe has large effects on individual refugees' psychological well-being, as well as on the healthcare systems of countries hosting refugees. For example, in Switzerland patients sometimes have to wait up to 12 months for the specific psychological treatment due to a lack of specialists. To address this problem the WHO has developed Problem Management Plus (PM+), a brief (five sessions), low-intensity psychological intervention, delivered by paraprofessionals, that addresses common mental disorders in people in communities affected by adversity. The effectiveness and implementation of PM+ has never been examined in Switzerland before, this is the aim of the current randomized controlled trial.

DETAILED DESCRIPTION:
Recent crises in the Middle East have resulted in an unprecedented increase in the worldwide number of refugees and asylum seekers. Switzerland (CH) is strongly affected by this crisis too.There are currently about 19'000 Syrian refugees and asylum seekers in Switzerland. A similar number of other Arabic-speaking individuals have applied for asylum in Switzerland since 2011. Due to the ongoing war in the MENA region, it is unlikely that this kind of migration and flight will resolve within the next years.

Refugees have typically been exposed to multiple stressors related to war and displacement including loss of family members, destruction of homes and livelihoods and human rights violations such as sexual violence or torture. They have often undertaken a risky and stressful flight leaving their homes for an unknown future. Accordingly, various studies have shown that refugees are at considerable risk of developing common mental disorders, including depression, anxiety, posttraumatic stress disorder (PTSD) and related somatic health symptoms.

According to the UNHCR, 85% of all displaced persons are hosted in third-world countries where appropriate mental health care is often not available. However, Western health systems are also often unable to appropriately cover the needs of this particularly vulnerable population regarding prevention and treatment of mental health problems. As a response to this situation, the WHO developed the low-intensity Problem Management Plus (PM+) programs, a new generation of short, resource-sparing, trans-diagnostic (i.e., not specifically aimed at treating a certain mental disorder) programs to reduce common mental health symptoms and improve psychosocial functioning. PM+ is based on the WHO treatment guidelines for conditions related to stress. PM+ is a 5-sessions intervention aimed at reducing symptoms of depression, anxiety, PTSD, and related conditions, is delivered by trained non-specialized workers or lay people, and is available in individual and group delivery formats for both children and adults. It comprises evidence-based techniques of (a) problem solving, (b) stress management, (c) behavioral activation, and (d) accessing social support. PM+ has been successfully tested for effectiveness in Kenya and Pakistan.

The STRENGTHS (Syrian REfuGees MeNTal HealTH Care Systems) study aims at evaluating the effectiveness and implementation of PM+ with Syrian refugees in different settings in low- and high-resource countries. The study consortium includes international experts in the domains of trauma and public mental health as well as representatives of WHO and UNHCR. The Zürich study site has been consigned to examine PM+ with adult refugees in an individual treatment setting in Switzerland. At the same time, similar studies in other countries will be undertaken. Despite the objective of these studies to implement and evaluate the effectiveness of PM+ in refugees, each research institution acts independently. Moreover, the other studies will be completed in different treatment settings - i.e., in children and adolescents (Lebanon), in groups (Turkey and Netherlands), and internet-delivered PM+ (Germany and Egypt).

To date, the effectiveness and implementation of PM+ has not been investigated in a highly industrialized country, such as Switzerland.

In the present study, the investigators will evaluate the effectiveness and implementation of PM+ in Arabic speaking refugees in Switzerland.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Arabic-speaking refugees or asylum seekers who entered Switzerland after March 2011
* ≥ 18 years of age
* Arabic-speaking (Levantine Arabic)
* Signed Informed Consent after being informed
* Increased psychological distress (K10 > 15)
* Reduced psychological functioning (WHODAS 2.0 > 16)

Exclusion Criteria:

* Inability to follow the procedures of the study
* Previous enrolment into the current study phase
* Participants under tutelage
* Acute or severe psychiatric (e.g. schizophrenia) or neurological illness (e.g. dementia)
* Imminent suicide risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in psychological distress | Baseline assessment, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment
  Change of psychological distress measured with the Hopkins Symptom Checklist (HSCL-25) serves as primary beneficiary-related health outcome. The 25 items are rated on a scale from 1 to 4. Higher scores indicate more pronounced symptom severity.

SECONDARY OUTCOMES:
Change in posttraumatic stress disorder symptoms | Baseline assessment, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment
  Change in posttraumatic stress disorder symptoms measured with the PTSD Checklist for DSM-5 (PCL-5). Responses are scored on a scale from 0 to 4 with higher scores indicating more pronounced symptom severity.
Change in functional disability | Screening, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment
  Change in functional disability measured with the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0). The items are rated on a scale from 1 to 5. Higher scores indicate more pronounced functional disability.

OTHER OUTCOMES:
Assessment of change in self-reported problems | Baseline assessment, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment
  Assessment of change in self-reported problems measured with the PSYCHLOPS. The Psychological Outcomes Profiles (PSYCHLOPS) scale is a patient-generated outcome measure, serving as an indicator of change in response to therapy. Items are rated on a scale from 1 to 5 (respectively 1 - 7) with lower scores indicating greater improvement in self reported problems.
Exposure to traumatic events | Measured at baseline assessment and 12-months follow up only
  Exposure to traumatic events will be assessed using the Traumatic Events (TE) - a combination of two standardized questionnaires, namely the Life Events Checklist and the Harvard Trauma Questionnaire.
Reduction of post-migration stressors | Baseline assessment, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment
  Changes in post-migration stressors will be assessed using a version of the Post-Migration Living Difficulties Checklist (PMLDC). Items are rated on a scale from 0 to 4 with lower scores representing fewer post-migration stressors.
Somatization and somatic symptoms | Baseline assessment, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment
  Somatization and somatic symptoms will be assessed using the Patient Health Questionnaire-15 (PHQ-15). Items are rated on a scale from 1 to 3. Higher scores indicate higher symptom severity.
Level of integration | Screening, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment
  Level of integration will be measured using the Immigration Policy Lab Integration Index (IPL-12).
General Self-Efficacy | Baseline assessment, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment
  General Self-Efficacy will be assessed using a short form of the General Self-Efficacy Scale (GSE-6). Reponses are given on a scale from 1 to 4 with higher scores representing higher general self-efficacy.
Attitudes towards mental health | Baseline assessment, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment
  Attitudes towards mental health will be measured with with a set of selected questions (e.g. "Mentally ill people tend to be violent").This questionnaire has been used with Syrian refugees in previous research.
Impact of COVID-19 pandemic | Baseline assessment, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment
  The impact of the COVID-19 pandemic will be assessed with a set of selected questions regarding medical state, psychological state, financial situation and resources (own questionnaire).
Cost of Care | Baseline assessment, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment
  The Client Service Receipt Inventory (CSRI) was developed for the collection of data on service utilization and related characteristics of people with mental disorders, as the basis for calculating the costs of care for mental health cost-effectiveness research.
Access to health care services | Baseline assessment
  A set of question regarding previous contact with the mental health care services and the previous experiences regarding the utilization of any forms of mental support (own questionnaire).
Assessing the extent to which the strategies taught in PM+ are used before and after the study participation with the Reducing Tension Checklist | Baseline assessment, 1 week post-intervention assessment (6 weeks after baseline), 3 month post-intervention assessment (4-4.5 months after baseline), 12 month post intervention assessment.
  The outcome is measured with a nine-item scale that was developed to assess the extent to which the participants perceives that they use the specific strategies, which are trained during the study intervention. The items are rated on a scale from 0 to 4. Higher scores represent greater usage of the strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Naser Morina, PhD, Principal Investigator — Klinik für Konsiliarpsychiatrie und Psychosomatik
Locations (1):
- Klinik für Konsiliarpsychiatrie und Psychosomatik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sijbrandij M, Acarturk C, Bird M, Bryant RA, Burchert S, Carswell K, de Jong J, Dinesen C, Dawson KS, El Chammay R, van Ittersum L, Jordans M, Knaevelsrud C, McDaid D, Miller K, Morina N, Park AL, Roberts B, van Son Y, Sondorp E, Pfaltz MC, Ruttenberg L, Schick M, Schnyder U, van Ommeren M, Ventevogel P, Weissbecker I, Weitz E, Wiedemann N, Whitney C, Cuijpers P. Strengthening mental health care systems for Syrian refugees in Europe and the Middle East: integrating scalable psychological interventions in eight countries. Eur J Psychotraumatol. 2017 Nov 7;8(sup2):1388102. doi: 10.1080/20008198.2017.1388102. eCollection 2017. PMID 29163867
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Background] Steel Z, Chey T, Silove D, Marnane C, Bryant RA, van Ommeren M. Association of torture and other potentially traumatic events with mental health outcomes among populations exposed to mass conflict and displacement: a systematic review and meta-analysis. JAMA. 2009 Aug 5;302(5):537-49. doi: 10.1001/jama.2009.1132. PMID 19654388
- [Background] Rahman A, Khan MN, Hamdani SU, Chiumento A, Akhtar P, Nazir H, Nisar A, Masood A, Din IU, Khan NA, Bryant RA, Dawson KS, Sijbrandij M, Wang D, van Ommeren M. Effectiveness of a brief group psychological intervention for women in a post-conflict setting in Pakistan: a single-blind, cluster, randomised controlled trial. Lancet. 2019 Apr 27;393(10182):1733-1744. doi: 10.1016/S0140-6736(18)32343-2. Epub 2019 Apr 1. PMID 30948286
- [Background] Bryant RA, Schafer A, Dawson KS, Anjuri D, Mulili C, Ndogoni L, Koyiet P, Sijbrandij M, Ulate J, Harper Shehadeh M, Hadzi-Pavlovic D, van Ommeren M. Effectiveness of a brief behavioural intervention on psychological distress among women with a history of gender-based violence in urban Kenya: A randomised clinical trial. PLoS Med. 2017 Aug 15;14(8):e1002371. doi: 10.1371/journal.pmed.1002371. eCollection 2017 Aug. PMID 28809935
- [Background] Fazel M, Wheeler J, Danesh J. Prevalence of serious mental disorder in 7000 refugees resettled in western countries: a systematic review. Lancet. 2005 Apr 9-15;365(9467):1309-14. doi: 10.1016/S0140-6736(05)61027-6. PMID 15823380
- [Background] Bogic M, Njoku A, Priebe S. Long-term mental health of war-refugees: a systematic literature review. BMC Int Health Hum Rights. 2015 Oct 28;15:29. doi: 10.1186/s12914-015-0064-9. PMID 26510473
- See also: Staatssekretariat für Migration. (2020a). Asylstatistik 2019. — https://www.sem.admin.ch/sem/de/home/publiservice/statistik/asylstatistik/archiv/2019.html
- See also: Staatssekretariat für Migration. (2020b). Asylstatistik (nach Nationen). — https://www.sem.admin.ch/sem/de/home/publiservice/statistik/asylstatistik/uebersichten.html
- See also: UNHCR (2020). Figures at a Glance. — https://www.unhcr.org/figures-at-a-glance.html